CLINICAL TRIAL: NCT02169817
Title: Bacillus Clausii in the Treatment of Acute Community-acquired Diarrhea Among Latin American Children (cadiLAc)
Brief Title: Evaluation Of Bacillus Clausii In Treatment Of Acute Diarrhea In Latin American Children
Acronym: cadiLAc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENTERR06929; U1111-1149-1704 (Other: UTN)
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Acute Gastroenteritis
MeSH Terms: interventions — clausin peptide, Bacillus clausii; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enterogermina + Enterolyte (Experimental): 2 vials of Enterogermina per day for 5 days and Enterolyte according to investigator´s recommendation
  Interventions: Drug: Bacillus clausii; Drug: Oral Rehydration Therapy

INTERVENTIONS:
Drug: Bacillus clausii — Pharmaceutical form:aqueous suspension Route of administration: oral
  Other Names: Enterogermina
Drug: Oral Rehydration Therapy — Pharmaceutical form:vials/sachets for solution Route of administration: oral
  Other Names: Enterolyte

SUMMARY:
Primary Objective:

To demonstrate the effectiveness of treatment with Bacillus clausii probiotic strain (Enterogermina) in combination with oral rehydration therapy (ORT) for a period of 5 days, in the duration of acute community-acquired diarrhea in Latin American children.

Secondary Objectives:

To evaluate the clinical safety of Enterogermina in acute diarrhea in children and to demonstrate its effectiveness on stool frequency, stool consistency, and number of vomiting episodes.

To evaluate parent's overall global assessment. To evaluate the safety and effectiveness of Enterogermina in norovirus acute gastroenteritis (AGE).

DETAILED DESCRIPTION:
The maximum duration of study participation for each patient can be 10 days.

ELIGIBILITY:
Inclusion criteria:

Infants or children with acute community-acquired diarrhea (≥3 liquid or watery stools occurring in a 24-hour period):

* with less than 48 hours duration
* aged between 6 months and 5 years of age
* whose parents or legal guardians have given their written informed consent
* with clinical indication for ORT per formula of World Health Organization

Exclusion criteria:

Infants or children with:

* presence of blood, pus, or mucus in stools
* severe dehydration
* untreatable vomiting
* antibiotics indication for the treatment of this acute diarrhea;
* hospitalization
* expected hospitalization for the next hours due to the poor clinical conditions
* treatment with antibiotics, probiotics, or prebiotics within a period of 2 weeks before enrolment (the use of probiotics and prebiotics in dairy food such as yoghurt, cheese, milk prior to the study is permitted)
* previous use (within 48 hours) of kaolin, pectin, bismuth subsalicylate, racecadotril, loperamide, atropine and other anticholinergic agents
* indication of any other ORT different from the one prescribed in the study
* chronic diseases including chronic diarrhea
* immunodeficiency (acquired or congenital immunodeficiency)
* other infectious comorbid conditions
* known hypersensitivity to Bacillus clausii (Enterogermina) or other probiotics
* parent/legal guardian who, in the opinion of the Investigator, is unable to complete the patient diary or bring the child for the follow-up visit
* participation in another clinical trial in the last 3 months prior to the start of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 629 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea-from the date and time of first intake of investigational product up to date and time of first appearance of a loose stool followed by two consecutive normal stools recorded in the patient diary | from Day 1 to Day 5

SECONDARY OUTCOMES:
Mean number of stools per day | Day 1 to Day 5
Effect on consistency of stool | Day 1 to Day 5
Number of vomiting episodes per day | Day 1 to Day 5
Parent / Legal guardian's assessment of children's overall acceptance of Enterogermina | Day 1 to Day 5
Parent / Legal guardian's assessment of children's overall general state | Day 1 to Day 5
Safety outcome: Adverse events collection reported by the parent / legal guardian in diary and checked by the investigator | Day 1 to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Argentina (3):
  - 04, Pilar, Buenos Aires
  - 01, Mar del Plata
  - 06, San Miguel de Tucumán
- Brazil (4):
  - 076002, Curitiba
  - 076006, Porto Alegre
  - 076003, Salvador
  - 076001, São Paulo
- 170002, Armenia, Colombia
- 484010, Mexico City, Mexico
- Peru (2):
  - 604001, Lima
  - 604003, Lima